CLINICAL TRIAL: NCT00869843
Title: Phase I Study of Saline Linked Monopolar Surface Radiofrequency (RF) Ablation of Hepatic Tumors
Brief Title: Study of Saline Linked Monopolar Surface Radiofrequency (RF) Ablation of Hepatic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-0343
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Malignant Liver Tumors; Liver Metastases From Colorectal Cancer
Keywords: Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group (Other)
  Interventions: Procedure: RF Ablation

INTERVENTIONS:
Procedure: RF Ablation

SUMMARY:
* To determine the depth of coagulation which is possible in human liver tissue using the saline linked RF Surface ablation with the Tissue Link floating ball.
* To determine the efficacy of the technique on surface liver tumors using saline linked RF surface ablati
* To determine a safe (non-popping upper limit) of power per area that will permit a 1 cm depth of tissue destruction without inflow occlusion an da 2 cm depth with inflow occlusion.

DETAILED DESCRIPTION:
Treatment Plan: Patients with resectable hepatic metastases confined to the liver and who are referred to the Study Chairs will undergo routine work-up for hepatic resection.

Operative Procedure:

Stage I will be completed and the data analyzed before Stage II commences. Stage I data will be used to define the safe levels for use in Stage II.

Stage I-Depth of coagulation with and without inflow occlusion at fixed times - and powers below the popping threshold.

At surgery, in the absence of extrahepatic disease, the liver will be dissected in the usual fashion for a bi-segmentectomy, hemihepatectomy or larger liver resection. Prior to transection of the liver, saline linked RF ablations will be performed on normal liver tissue within the area of resection away from the tumor and the proposed line of transection.

1 cm and 2 cm diameters will be studied together in 8 patients. They will be treated for a total of 18 minutes (9 min for 1 cm and 9 min for 2 cm with 9 minutes of inflow occlusion. The 4 cm lesions will be studied in 8 other patients, 4 of whom will receive 9 minutes of inflow occlusion.

After resection of the liver and establishment of resection margins on the tumor, the ablated areas of normal liver tissue will be excised frozen and studied for depth of lesion and examined by H & E and histological techniques using vital stains that will allow definition of tissue depth.

Stage II-An ablate and resect Study

Once parameters have been defined on normal liver, the effect of surface RF ablation on resectable hepatic tumors which come to the surface of the liver will be examined. In this portion of the study, tumors will be treated with saline linked RF ablation with a power and a duration of application which has been found to produce the maximum safe depth of coagulation. The surface area of coagulation will be dependent upon the size of the tumor. The area of treatment will encompass the tumor as well as a zone at least 0.5cm outside the edge of the tumor. Inflow occlusion will be used in one half of the patients.

After resection of the liver and establishment of resection margins on the tumor, the ablated areas will be excised frozen and studied for depth of lesion and examined by H & E and histological techniques using vital stains that will allow definition of tissue depth. Twelve tumors will be treated in 12 patients.

Pathology Evaluation

First Group of Patients The normal tissue exposed to RF will be resected, prepared for histo-pathological studies and examined to determine the extent of tissue necrosis and popping, if any.

Second Group of Patients Tumors exposed to RF ablation will be resected and the extent of tissue necrosis and popping will be determined. Also, damage to normal tissue will be examined.

ELIGIBILITY:
Eligibility for Stage I (Normal Liver Tissue)

* Resectable liver metastases from malignant liver tumors, primary or secondary
* Patient has been scheduled for liver resection and is in generally good medical condition
* No evidence of extra-hepatic disease
* Patient does not have a pacemaker
* Age >= 18
* Able to provide informed consent

Eligibility for Stage II (Patients with liver metastases from colorectal cancer)

* Resectable liver metastases from colorectal cancer
* Patient has been scheduled for liver resection is in generally good medical condition
* No evidence of extra-hepatic disease.
* Patient does not have a pacemaker
* Age >= 18
* Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-10; Primary Completion 2007-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Depth of coagulation which is possible in human liver tissue using the saline linked RF Surface ablation with the Tissue Link floating ball | Day 1
  On day of surgery
Efficacy of the technique on surface liver tumors using saline lined RF Surface ablation. | Day 1
  On day of surgery

SECONDARY OUTCOMES:
Determine a safe (non-popping upper limit) of power per area that will permit a 1 cm depth of tissue destruction without inflow occlusion and a 2 cm depth with inflow occlusion. | Day 1
  On day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Steven Strasberg, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Gnerlich JL, Ritter JH, Linehan DC, Hawkins WG, Strasberg SM. Saline-linked surface radiofrequency ablation: a safe and effective method of surface ablation of hepatic metastatic colorectal cancer. Ann Surg. 2009 Jul;250(1):96-102. doi: 10.1097/SLA.0b013e3181ae91af. PMID 19561459
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu